CLINICAL TRIAL: NCT01111071
Title: Variation Between Hospitals in Short-term Mortality After Acute Coronary Syndromes: A CALIBER Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Barts & The London NHS Trust (Other); Queen Mary University of London (Other); University of Bristol (Other); Yale University (Other)
Responsible Party: Principal Investigator, Julie George, NIHR Doctoral Fellow, University College, London
Other Study IDs: CALIBER-09-03; RP-PG-0407-10314 (Other Grant/Funding Number: National Institute of Health Research (UK))
Record Dates: First submitted 2010-04-16; First posted 2010-04-27 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Acute Coronary Syndrome
Keywords: hospital variation; 30 day mortality; in hospital mortality; acute coronary syndrome; myocardial infarction; unstable angina; hospital performance; trends
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- STEMI: patients with discharge diagnosis of ST elevation myocardial infarction
- nSTEMI: patients with discharge diagnosis of non ST elevation myocardial infarction
- unstable angina: patients with discharge diagnosis of unstable angina

SUMMARY:
We seek to investigate whether hospitals in England and Wales vary in their rate of mortality following admission for heart attack or unstable angina, the extent of such variation, whether discharge diagnosis affects the extent of variation, and whether such variation has changed over time. Furthermore, we will investigate what individual- or hospital-level factors explain variation in mortality between hospitals.

DETAILED DESCRIPTION:
Several studies have looked at between-hospital variation in mortality following myocardial infarction but have lacked patient-level data. Those with individual-level data have been limited by:

* use of in-hospital mortality as an outcome measure, which can be affected by length of stay,
* restriction to patients aged 65 and over, or otherwise selected patients, and
* patient-level explanatory factors lacking clinical detail, particularly medications given in hospital.

MINAP patient-level data allow the investigation of hospital variation in mortality (in-hospital and 30-day) in a group of unselected patients, taking into account clinical details such as medication use in hospital, as well as features of the hospitals providing care. The proposed study will establish the extent of variation between hospitals in England and Wales, whether this varies by ACS diagnosis, whether the variation has reduced over time and finally which patient-level or hospital-level factors explain any variation found.

A statistical analytic protocol for this study, dated 15.4.2010, is available on request.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* admitted between January 2003 to June 2009 (or latest date data available)

Exclusion Criteria:

* admitted to hospital with fewer than 25 admissions in given year

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with acute coronary syndrome to acute hospitals in England and Wales participating in the Myocardial Ischaemia National Audit Project (MINAP)
Sampling Method: Non-Probability Sample
Enrollment: 316648 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
all-cause 30-day mortality | 30 day
  all-cause 30-day mortality following hospitalisation for acute coronary syndrome

SECONDARY OUTCOMES:
all-cause in-hospital mortality | length of hospital stay
  all-cause in-hospital mortality following hospitalisation for acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Julie L George, MSc, Principal Investigator — University College, London
Locations (1):
- Epidemiology and Public Health, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
permissions to use anonymised data from data owners do not allow further sharing.

REFERENCES:
- [Background] Bradley EH, Herrin J, Elbel B, McNamara RL, Magid DJ, Nallamothu BK, Wang Y, Normand SL, Spertus JA, Krumholz HM. Hospital quality for acute myocardial infarction: correlation among process measures and relationship with short-term mortality. JAMA. 2006 Jul 5;296(1):72-8. doi: 10.1001/jama.296.1.72. PMID 16820549
- [Background] Heidenreich PA, Lewis WR, LaBresh KA, Schwamm LH, Fonarow GC. Hospital performance recognition with the Get With The Guidelines Program and mortality for acute myocardial infarction and heart failure. Am Heart J. 2009 Oct;158(4):546-53. doi: 10.1016/j.ahj.2009.07.031. PMID 19781413
- [Background] Peterson ED, Roe MT, Mulgund J, DeLong ER, Lytle BL, Brindis RG, Smith SC Jr, Pollack CV Jr, Newby LK, Harrington RA, Gibler WB, Ohman EM. Association between hospital process performance and outcomes among patients with acute coronary syndromes. JAMA. 2006 Apr 26;295(16):1912-20. doi: 10.1001/jama.295.16.1912. PMID 16639050
- [Background] Alter DA, Austin PC, Tu JV; Canadian Cardiovascular Outcomes Research Team. Community factors, hospital characteristics and inter-regional outcome variations following acute myocardial infarction in Canada. Can J Cardiol. 2005 Mar;21(3):247-55. PMID 15776114
- [Background] Krumholz HM, Chen J, Wang Y, Radford MJ, Chen YT, Marciniak TA. Comparing AMI mortality among hospitals in patients 65 years of age and older: evaluating methods of risk adjustment. Circulation. 1999 Jun 15;99(23):2986-92. doi: 10.1161/01.cir.99.23.2986. PMID 10368115
- [Background] Krumholz HM, Wang Y, Mattera JA, Wang Y, Han LF, Ingber MJ, Roman S, Normand SL. An administrative claims model suitable for profiling hospital performance based on 30-day mortality rates among patients with an acute myocardial infarction. Circulation. 2006 Apr 4;113(13):1683-92. doi: 10.1161/CIRCULATIONAHA.105.611186. Epub 2006 Mar 20. PMID 16549637
- [Background] Krumholz HM, Wang Y, Chen J, Drye EE, Spertus JA, Ross JS, Curtis JP, Nallamothu BK, Lichtman JH, Havranek EP, Masoudi FA, Radford MJ, Han LF, Rapp MT, Straube BM, Normand SL. Reduction in acute myocardial infarction mortality in the United States: risk-standardized mortality rates from 1995-2006. JAMA. 2009 Aug 19;302(7):767-73. doi: 10.1001/jama.2009.1178. PMID 19690309
- [Background] Granger CB, Steg PG, Peterson E, Lopez-Sendon J, Van de Werf F, Kline-Rogers E, Allegrone J, Dabbous OH, Klein W, Fox KA, Eagle KA; GRACE Investigators. Medication performance measures and mortality following acute coronary syndromes. Am J Med. 2005 Aug;118(8):858-65. doi: 10.1016/j.amjmed.2005.01.070. PMID 16084178
- [Background] Rasmussen S, Zwisler AD, Abildstrom SZ, Madsen JK, Madsen M. Hospital variation in mortality after first acute myocardial infarction in Denmark from 1995 to 2002: lower short-term and 1-year mortality in high-volume and specialized hospitals. Med Care. 2005 Oct;43(10):970-8. doi: 10.1097/01.mlr.0000178195.07110.d3. PMID 16166866
- [Background] Rasmussen S, Abildstrom SZ, Rasmussen JN, Gislason GH, Schramm TK, Folke F, Kober L, Torp-Pedersen C, Madsen M. Hospital variation in use of secondary preventive medicine after discharge for first acute myocardial infarction during 1995-2004. Med Care. 2008 Jan;46(1):70-7. doi: 10.1097/MLR.0b013e3181484952. PMID 18162858
- [Background] Rosato S, Seccareccia F, D'Errigo P, Fusco D, Maraschini A, Badoni G, Perucci CA. Thirty-day mortality after AMI: effect modification by gender in outcome studies. Eur J Public Health. 2010 Aug;20(4):397-402. doi: 10.1093/eurpub/ckp194. Epub 2009 Nov 27. PMID 19946045
- [Background] Popescu I, Werner RM, Vaughan-Sarrazin MS, Cram P. Characteristics and outcomes of America's lowest-performing hospitals: an analysis of acute myocardial infarction hospital care in the United States. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):221-7. doi: 10.1161/CIRCOUTCOMES.108.813790. Epub 2009 May 5. PMID 20031841
- [Background] Kosseim M, Mayo NE, Scott S, Hanley JA, Brophy J, Gagnon B, Pilote L. Ranking hospitals according to acute myocardial infarction mortality: should transfers be included? Med Care. 2006 Jul;44(7):664-70. doi: 10.1097/01.mlr.0000215848.87202.c7. PMID 16799361
- [Background] Murphy NF, MacIntyre K, Stewart S, Capewell S, McMurray JJ. Reduced between-hospital variation in short term survival after acute myocardial infarction: the result of improved cardiac care? Heart. 2005 Jun;91(6):726-30. doi: 10.1136/hrt.2004.042929. PMID 15894761
- [Background] Leyland AH, Boddy FA. League tables and acute myocardial infarction. Lancet. 1998 Feb 21;351(9102):555-8. doi: 10.1016/S0140-6736(97)09362-8. PMID 9492774
- See also: CArdiovascular disease research Linking Bespoke studies and Electronic Records — http://www.caliberresearch.org